CLINICAL TRIAL: NCT00262080
Title: A Double-blind, Placebo-controlled Study (72 Patients, Randomized 1:1) Followed by a Repeat-dosing Phase to Assess the Efficacy and Safety of DX-88 (Ecallantide; Recombinant Plasma Kallikrein Inhibitor) for the Treatment of Acute Attacks of Hereditary Angioedema
Brief Title: Efficacy and Safety Study of DX-88 to Treat Acute Attacks of Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDEMA3 (DX-88/14)
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Results first posted 2010-05-11 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — ecallantide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DX-88 (ecallantide) (Experimental): DX-88 (ecallantide) 30 mg given as three 10 mg/mL subcutaneous injections.
  Interventions: Drug: ecallantide
- Placebo (Placebo Comparator): Phosphate Buffer Saline (PBS), pH 7.0 given as 3 subcutaneous injections.
  Interventions: Drug: Phosphate Buffer Saline (PBS),

INTERVENTIONS:
Drug: ecallantide — dose of 30 mg (10 mg/ml) given as 3 subcutaneous injections.
  Other Names: DX-88
  Arms: DX-88 (ecallantide)
Drug: Phosphate Buffer Saline (PBS), — given as three 1mL subcutaneous injections.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a subcutaneous dose of DX-88 (ecallantide; an investigational product) is safe and relieves symptoms of HAE in patients suffering from moderate to severe acute attacks of HAE.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 and older
* Documented diagnosis of HAE, Type I or II
* Executed informed consent
* Presentation for treatment within 8 hours of patient recognition of moderate to severe HAE attack

Exclusion Criteria:

* Receipt of investigational drug or device, other than DX-88, within 30 days of treatment
* Receipt of non-investigational C1-INH (C1 esterase inhibitor) within 7 days of treatment
* Diagnostic of acquired angioedema, estrogen-dependent angioedema or drug induced angioedema
* Pregnancy or breastfeeding
* Patients who have received DX-88 within 7 days of presentation for dosing in the Double-blind Phase

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2005-12-31 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2007-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Institute for Asthma and Allergy, Wheaton, Maryland, United States

REFERENCES:
- [Derived] Rubinstein E, Stolz LE, Sheffer AL, Stevens C, Bousvaros A. Abdominal attacks and treatment in hereditary angioedema with C1-inhibitor deficiency. BMC Gastroenterol. 2014 Apr 9;14:71. doi: 10.1186/1471-230X-14-71. PMID 24712435
- [Derived] MacGinnitie AJ, Davis-Lorton M, Stolz LE, Tachdjian R. Use of ecallantide in pediatric hereditary angioedema. Pediatrics. 2013 Aug;132(2):e490-7. doi: 10.1542/peds.2013-0646. Epub 2013 Jul 22. PMID 23878046
- [Derived] Sheffer AL, MacGinnitie AJ, Campion M, Stolz LE, Pullman WE. Outcomes after ecallantide treatment of laryngeal hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2013 Mar;110(3):184-188.e2. doi: 10.1016/j.anai.2012.12.007. Epub 2013 Jan 5. PMID 23548529
- [Derived] Bernstein JA, Shea EP, Koester J, Iarrobino R, Pullman WE. Assessment of rebound and relapse following ecallantide treatment for acute attacks of hereditary angioedema. Allergy. 2012 Sep;67(9):1173-80. doi: 10.1111/j.1398-9995.2012.02864.x. Epub 2012 Jul 5. PMID 22765833
- [Derived] Riedl M, Campion M, Horn PT, Pullman WE. Response time for ecallantide treatment of acute hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2010 Dec;105(6):430-436.e2. doi: 10.1016/j.anai.2010.09.005. Epub 2010 Oct 25. PMID 21130380
- [Derived] Cicardi M, Levy RJ, McNeil DL, Li HH, Sheffer AL, Campion M, Horn PT, Pullman WE. Ecallantide for the treatment of acute attacks in hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):523-31. doi: 10.1056/NEJMoa0905079. PMID 20818887

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were screened in advance of presenting with an Hereditary Angioedema (HAE) attack but were randomized only upon attack.
Groups:
- Ecallantide / Ecallantide: Patients treated with ecallantide in the double-blind part and eligible for treatment with ecallantide in the repeat-dosing part of the study once their Follow-up Visit 1 (Day 7) in the double-blind part was completed.
- Placebo / Ecallantide: Patients treated with placebo in the double-blind part and eligible for treatment with ecallantide in the repeat-dosing part of the study once their Follow-up Visit 1 (Day 7) in the double-blind part was completed.
- Ecallantide (Repeat Dose Only): Patients not treated in the double-blind part but treated with ecallantide in the repeat-dosing part.
Period: Double Blind Treatment Period
Arm/Group | Ecallantide / Ecallantide | Placebo / Ecallantide | Ecallantide (Repeat Dose Only)
Started | 36 (One patient was randomized to receive ecallantide but was treated with placebo.) | 36 (One patient was randomized to receive placebo but was treated with ecallantide.) | 0
Completed | 35 | 36 | 0
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Repeat Dose Treatment Period
Arm/Group | Ecallantide / Ecallantide | Placebo / Ecallantide | Ecallantide (Repeat Dose Only)
Started | 22 (Not all patients treated in the double-blind part came for treatment in the repeat-dose part.) | 26 (Not all patients treated in the double-blind part came for treatment in the repeat-dose part.) | 19 (This arm represents new patients, not treated in the double-blind part of the study.)
Completed | 18 (Some patients participated in only the double-blind or the open label phase.) | 25 | 14
Not Completed | 4 | 1 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Decision to discontinue the study | 0 | 0 | 2
Not completed — enrolled in EDEMA4 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ecallantide / Ecallantide: Patients treated with ecallantide in the double-blind part (ITT as treated) and eligible for treatment with ecallantide in the repeat-dosing part of the study once their Follow-up Visit 1 (Day 7) in the double-blind part was completed.
- Placebo / Ecallantide: Patients treated with placebo in the double-blind part (ITT as treated) and eligible for treatment with ecallantide in the repeat-dosing part of the study once their Follow-up Visit 1 (Day 7) in the double-blind part was completed.
- Ecallantide (Repeat-Dosing Part Only): Patients not treated in the double-blind part but treated with ecallantide in the repeat-dosing part. One patient was omitted from analysis in the intent-to-treat and per-protocol populations due to the loss of the data for the 4-hour post-dose assessments during treatment episode 1.
- Total: Total of all reporting groups
Arm/Group | Ecallantide / Ecallantide | Placebo / Ecallantide | Ecallantide (Repeat-Dosing Part Only) | Total
Number analyzed (Participants) | 36 | 36 | 18 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (14.3) | 33.6 (14.6) | 35.0 (14.6) | 34.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 11 | 58
  Male | 13 | 12 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Treatment Outcome Score at 4 Hours Post-Dose
Description: Treatment Outcome Score (TOS) is a validated, comprehensive measure of symptom response to treatment. At 4 hours , patient assessment of response characterized by their change from baseline in symptom severity and collected by anatomic site of attack involvement, was recorded on a categorical scale (significant improvement [100] to significant worsening [-100]). The response at each anatomic site was weighted by baseline severity and then the weighted scores across all involved sites were averaged to calculate the TOS. Clinically meaningful improvement was indicated by a TOS of 30 or higher.
Time Frame: 4 hours post-dose (DOUBLE-BLIND PART)
Population: ITT as treated: two patients randomized on the same day at the same study center were administered treatment opposite to their randomized treatment assignment. Data were analyzed based on actual treatment received. Imputation was used to account for emerging symptoms and medical intervention. Best possible score = 100; worst possible score = -100.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ecallantide: Patients treated with ecallantide in the double-blind part.
- Placebo: Patients treated with placebo in the double-blind part.
Arm/Group | Ecallantide | Placebo
Number analyzed (Participants) | 36 | 36
units on a scale | 49.5 (59.43) [50 to 100] | 18.5 (67.78) [75 to 100]
Statistical Analysis 1: Comparison: Ecallantide vs Placebo; The primary efficacy analysis compared the TOS at 4 hours post-dosing for patients treated with ecallantide and placebo. Treatment effect was assessed by the non-parametric Wilcoxon Rank Sum test because of an assumed non-normal distribution; Test type: Superiority or Other; p = 0.037, non-parametric Wilcoxon Rank Sum test — no adjustment was made for multiple comparisons. Treatment effect will be deemed statistically significant if the coefficient for the treatment group within the statistical model is significant at level 0.05

2. Secondary Outcome: Change From Baseline in Mean Symptom Complex Severity (MSCS) Score at 4 Hours Post-dose
Description: Mean Symptom Complex Severity (MSCS) score is a validated, comprehensive point-in-time measure of symptom severity. At baseline and 4 hours, patients rated the severity on a categorical scale (0 = normal, 1 = mild, 2 = moderate, 3 = severe) for symptoms at each affected anatomical location. Ratings were averaged to obtain the MSCS score. A decrease in MSCS score reflected an improvement in symptoms; clinically meaningful improvement (minimally important difference) was indicated by a reduction in the score of 0.30 or more.
Time Frame: baseline, 4 hours post-dose (DOUBLE-BLIND PART)
Population: ITT as treated: two patients randomized on the same day at the same center were administered treatment opposite to their randomized treatment assignments. Data were analyzed based on their actual treatment received. Imputation was used to account for emerging symptoms and medical intervention. Best possible score = 0.0; worst possible score = 3.0.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ecallantide | Placebo
Number analyzed (Participants) | 36 | 36
units on a scale
  MSCS Score at baseline | 2.17 (0.51) | 2.24 (0.55)
  MSCS Score at 4 hours post-dose | 1.26 (0.96) | 1.75 (0.90)
  Change from baseline in MSCS at 4 hours post-dose | -0.91 (1.10) | -0.48 (0.68)
Statistical Analysis 1: Comparison: Ecallantide vs Placebo; The analysis compared the change from baseline in MSCS score at 4 hours post-dosing for patients treated with ecallantide and placebo. Treatment effect was assessed by the non-parametric Wilcoxon Rank Sum test because of an assumed non-normal distribution; Test type: Superiority or Other; p = 0.044, Wilcoxon Rank Sum Test. — [p-value comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Number of Patients With Symptom Complexes of Treated Attack at Baseline(DOUBLE-BLIND PART)
Description: Patient-reported severity of symptom complexes at baseline, by symptom complex and treatment group. Patients were to have at least one symptom complex that was moderate or severe. Patients could present with multiple symptom complexes, some of which could be mild. Mild=noticeable but do not impact daily living activities; Moderate=treatment or intervention is highly desirable and activities of daily living are impacted; Severe=require treatment or intervention due to inability to perform activities of daily living. The results are for number of patients with symptom complexes including mild, moderate and severe, provided the patients have at least one symptom complex that was moderate or severe
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Ecallantide | Placebo
Number analyzed (Participants) | 36 | 36
participants
  Internal Head/Neck Symptoms | 9 | 4
  Stomach/GI | 19 | 22
  Genital/Buttocks | 2 | 4
  External Head/Neck | 5 | 8
  Cutaneous | 21 | 14

4. Other Pre Specified Outcome: Treatment Outcome Score at 4 Hours Post-Dose Over Multiple Treatment Episodes
Description: as for outcome 1
Time Frame: 4 hours post-dose (REPEAT-DOSING PART)
Population: Treatment episode 1 contains data only from those participants who were new patients in the repeat-dosing part. Treatment episode 2 and beyond contain data pooled from patients treated in the double-blind part (ecallantide or placebo) and the repeat-dosing part. Data imputation was used to account for emerging symptoms and medical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ecallantide: Patients treated with ecallantide in the repeat-dose part.
Arm/Group | Ecallantide
Number analyzed (Participants) | 51
units on a scale
  Episode 1 (n =18) | 71.3 (28.85)
  Episode 2 (n = 51) | 73.3 (44.9)
  Episode 3 (n = 30) | 81.9 (28.52)
  Episode 4 (n = 21) | 81.2 (24.53)
  Episode 5 (n = 11) | 48.5 (68.5)
  Episode 6 (n = 9) | 60.4 (49.26)

5. Other Pre Specified Outcome: Change From Baseline in Mean Symptom Complex Severity (MSCS) Score at 4 Hours Post-dose Over Multiple Treatment Episodes
Description: The Mean Symptom Complex Severity (MSCS) score is a validated, comprehensive point-in-time measure of symptom severity. At baseline and 4 hours, patients rated the severity on a categorical scale (0 = normal, 1 = mild, 2 = moderate, 3 = severe) for symptoms at each affected anatomical location. Ratings were averaged to obtain the MSCS score. A decrease in MSCS score reflected an improvement in symptoms; clinically meaningful improvement was indicated by a reduction in the score of 0.30 or more.
Time Frame: baseline, 4 hours post-dose (REPEAT-DOSING PART)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ecallantide
Number analyzed (Participants) | 51
units on a scale
  Episode 1 (n = 17) | -1.16 (0.87)
  Episode 2 (n = 51) | -1.12 (0.90)
  Episode 3 (n = 30) | -1.31 (0.87)
  Episode 4 (n = 21) | -1.38 (0.79)
  Episode 5 (n = 11) | -0.89 (0.72)
  Episode 6 (n = 9) | -0.87 (0.75)

6. Secondary Outcome: Time to Significant Improvement in Overall Response
Description: The overall response assessment is a patient-reported assessment of global response to therapy. Patients are asked to perform an overall response assessment at regular intervals, relative to baseline. Patients were asked "overall how are you feeling" compared to how they felt before study drug. Answer options were "a lot worse", "a little worse", "same", "a little better" or "a lot better or resolved". Significant improvement was the first time that the patient responded to the assessment as "a little better or resolved".
Time Frame: 4 hours post-dose (DOUBLE-BLIND PART)
Population: ITT as treated. Patients not reporting significant improvement before 4 hours were censored at 4 hours. Patients receiving additional HAE therapy within 4 hours were censored at the time of the medical intervention. The time to significant improvement is not provided in this display as the median time for placebo was not reached by 4 hours.
Measure: Number; unit: participant
Arm/Group | Ecallantide | Placebo
Number analyzed (Participants) | 36 | 36
participant
  Patients with Significant Improvement | 19 | 11
  Patients with Censored Data | 17 | 25
Statistical Analysis 1: Comparison: Ecallantide vs Placebo; The Log-Rank test was used to compare the time distribution between the two treatment groups; Test type: Superiority or Other; p = 0.055, Log Rank — [p-value comment as in outcome 1, analysis 1]

7. Other Pre Specified Outcome: Time to Significant Improvement in Overall Response Over Multiple Treatment Episodes
Description: The overall response assessment is a patient-reported assessment of global response to therapy. Patients are asked to perform an overall response assessment at regular intervals, relative to baseline (ie,immediately before treatment) using the following 5-category scale from significant improvement (Score = 100)to significant worsening (Score = -100)
Time Frame: 4 hours post-dose (REPEAT-DOSING PART)
Population: Patients not reporting significant improvement before 4 hours were censored at 4 hours. Patients receiving additional HAE therapy within 4 hours were censored at the time of the medical intervention. The time to significant improvement is not provided in this display as the interquartile range (IQR) was not reached by 4 hours for most episodes.
Measure: Number; unit: participants
Arm/Group | Ecallantide
Number analyzed (Participants) | 51
participants
  Episode 1 (n=18) | 10
  Episode 2 (n=51) | 37
  Episode 3 (n=30) | 24
  Episode 4 (n=21) | 14
  Episode 5 (n=11) | 6
  Episode 6 (n=9) | 5

ADVERSE EVENTS:
Time Frame: Adverse events were reported from enrollment (Study Day 1) through the conclusion of the Follow-up Visit 2 (Study Days 23-37) of each episode.
Description: Additionally, AEs suspected to be related to study procedures were collected from the time of informed consent through enrollment and from Follow-up Visit 2 through Follow-up Visit 3 (Study Days 83-97).
Groups:
- Double Blind - Ecallantide: Patients treated with ecallantide in the double-blind part only.
- Double-Blind Placebo: Patients treated with placebo in the double-blind part only.
- Repeat-Dosing Ecallantide: All patients treated with ecallantide in the repeat-dosing part, regardless of whether they were treated previously in the double-blind part or not. All adverse events reported in all repeat-dosing episodes are included. Patients reporting more than 1 AE with the same preferred term are counted only once for that preferred term.
Arm/Group | Double Blind - Ecallantide | Double-Blind Placebo | Repeat-Dosing Ecallantide
Serious Adverse Events (participants affected / at risk) | 3/36 | 2/36 | 7/67
Other Adverse Events (participants affected / at risk) | 13/36 | 7/36 | 22/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind - Ecallantide (N=36) | Double-Blind Placebo (N=36) | Repeat-Dosing Ecallantide (N=67)
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea Infectious (Infections and infestations) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Hereditary Angioedema (Congenital, familial and genetic disorders) | 3 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lymphoproliferative disorders (Blood and lymphatic system disorders) | 0 | 0 | 1
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash Generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind - Ecallantide (N=36) | Double-Blind Placebo (N=36) | Repeat-Dosing Ecallantide (N=67)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3
Headache (Nervous system disorders) | 4 | 2 | 10
Hereditary Angioedema (Congenital, familial and genetic disorders) | 0 | 2 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 0 | 6
Prothrombin Time Prolonged (Investigations) | 0 | 2 | 1
Pyrexia (General disorders) | 3 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dyax agreements vary, but Dyax will not prohibit any investigator from publishing. Dyax reviews publications prior to public release and can request deferral by up to 60 days beyond the proposed publication date if necessary to preserve its intellectual property. Dyax can request changes to publications to remove non-study-related confidential information. Dyax can also request deferral of single-center publications until after disclosure of the clinical trial's primary publication.